CLINICAL TRIAL: NCT07201857
Title: Peri-habilitation to Enhance Treatment Outcomes and Postoperative Recovery in Patients With Gastric Cancer
Brief Title: Peri-habilitation for Patients With Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University (Other)
Responsible Party: Principal Investigator, Min, Jae-Seok, Assistant Professor of Surgery, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KUMCANAM2025GES1
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer (Diagnosis); Gastric Cancer Patient; Gastric Cancer Patients Undergoing Gastrectomy; Gastric Cancer Patients Undergoing Minimally Invasive Gastrectomy; Gastric Cancer Patients Undergoing Laparoscopic Gastrectomy
Keywords: peri-habilitation; gastric cancer; postoperative recovery; exercise intervention
MeSH Terms: conditions — Stomach Neoplasms; Disease | interventions — Nutrition Assessment; Nutritional Status; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition (NUT) (Active Comparator): Nutrition (NUT) Participants will receive standard clinical care combined with nutrition education and protein-enriched soy milk supplementation for approximately 2 weeks before surgery and about 3 weeks after hospital discharge.
  Interventions: Dietary Supplement: nutrition education plus active supplement
- Exercise and Nutrition(EN) (Experimental): Exercise and Nutrition Group (EN)
  Participants will receive peri-habilitation exercise training in combination with nutritional intervention, including carbohydrate plus protein-enriched soy milk supplementation twice daily (before and after exercise), for approximately 2 weeks before surgery and about 3 weeks after hospital discharge.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: nutrition education plus active supplement — Nutrition Group (NUT) Participants will receive standard clinical care combined with nutrition education and protein-enriched soy milk supplementation for approximately 2 weeks before surgery and about 3 weeks after hospital discharge.
  Other Names: Nutrition
  Arms: Nutrition (NUT)
Behavioral: Exercise — Exercise and Nutrition
  Participants will receive peri-habilitation exercise training together with nutritional intervention, including carbohydrate plus protein-enriched soy milk supplementation twice daily (before and after exercise), for approximately 2 weeks before surgery and about 3 weeks after hospital discharge.
  Other Names: Exercise and Nutrition
  Arms: Exercise and Nutrition(EN)

SUMMARY:
This study aims to evaluate the clinical applicability of a peri-habilitation program in patients with gastric cancer by applying nutritional intervention for approximately two weeks before surgery and a combined exercise and nutrition intervention for about three weeks after hospital discharge, and by analyzing its effects on the prevention of postoperative complications and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older who have been diagnosed with gastric cancer and are scheduled to undergo surgical treatment or chemotherapy.

Exclusion Criteria:

* Patients with severe conditions who are unable to undergo the intervention prior to surgical treatment or chemotherapy.
* Patients with physical (e.g., musculoskeletal) or mental disorders that make participation in or continuation of the program impossible.
* Patients judged to be at risk of additional physical burden from the intervention.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed test | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Time to walk 4 meters (or 3 meters) at a normal, comfortable pace.
  * Seconds(sec)
  * Lower values(seconds) indicate better performance (faster walking speed)
Chair stand test | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Time to stand up and sit down 5 times from a chair without using the arms.
  * Seconds(sec)
  * Lower values(seconds) indicate better performance.
Balance test | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Time maintaining balance in three positions (feet together, semi-tandem, and tandem stance). The maximum time allowed for each position is 10 seconds.
  * Seconds(sec)
  * Higher values(seconds) indicate better performance.
Timed up and go test | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Time to stand up from a chair, walk 3 meters, turn around, walk back, and sit down.
  * Seconds(sec)
  * Lower values(seconds) indicate better performance.

SECONDARY OUTCOMES:
Electrocardiogram(ECG) | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Cardiovascular status assessed using electrocardiogram (ECG)
  * N/A (qualitative/clinical assessment)
  * Abnormal ECG findings indicate impaired cardiovascular function.
Inflammation and Oxidative Stress Markers (Blood Analysis) | Baseline (2 weeks before surgery) Preoperative hospitalization (1-4 days before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Inflammatory and oxidative stress markers assessed by blood analysis, including C-reactive protein (CRP) and white blood cell(WBC) count.
  * mg/L for CRP; ×10⁹/L for WBC
  * Higher values indicate greater systemic inflammation.
Hospital Anxiety and Depression Scale (HADS) | Baseline (2 weeks before surgery) Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * The scale ranges from 0 to 21 points for each domain (anxiety and depression). Higher scores indicate worse psychological distress.
  * Score on a scale (0-21)
  * Higher scores indicate worse psychological condition.
Quality of life(KOQUSS-32, KOQUSS-40) | Baseline (2 weeks before surgery) 3 weeks after discharge 6 months after surgery
  * Quality of life assessed using the Korean Quality of Life in Stomach Cancer Patient Study group questionnaires (KOQUSS-32 and KOQUSS-40). Each questionnaire provides domain-specific scores. Higher scores indicate better quality of life.
  * Score on a scale (range depends on quetionnaire)
  * Higher scores indicate better quality of life.
Clavien-dindo classification | Postoperative discharge (at hospital discharge) 3 weeks after discharge 6 months after surgery
  * Postoperative complications will be assessed and graded according to the Clavien-Dindo classification system (Grade I-V).
  * Number of participants with each complication grade.
  * Higher grades indicate more severe postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Anam Hospital, Seoul, seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided